CLINICAL TRIAL: NCT00284895
Title: The Effect of Medical and Surgical Weight Loss on Pulmonary Physiology and Airway
Brief Title: The Effect of Obesity on Lung Functioning
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Other Study IDs: NJC HS1963
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Obesity; Asthma
Keywords: Obesity; Bariatric Surgery; Weight Loss Surgery; Asthma
MeSH Terms: conditions — Obesity; Asthma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This research study is looking at the effects of weight loss, due to surgery or structured weight-loss program on lung function, inflammation in your body and lungs, asthma and asthma symptoms. This study is important because we will be better able to understand the effect of weight on lung functioning and asthma. Approximately 20 research subjects will be enrolling in this study at National Jewish.

Adults with asthma who has elected to undergo weight-reduction surgery may qualify for the participation. Involvement will last about 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18yr) who report a physician's diagnosis of asthma and have taken any asthma medication within the last 2 weeks.
* Obesity (Body Mass Index (BMI) ≥40, or ≥35 with comorbidities, as per published guidelines for qualification for bariatric surgery).
* Planned weight-loss surgery or structured weight-loss plan.

Exclusion Criteria:

* Tobacco use within one month.
* Qualifying lung-functioning.
* Qualifying oxygen saturation levels.
* Use of systemic corticosteroids (Prednisone) within one month.
* Presence of another chronic lung disease besides asthma (COPD, bronchiectasis, ILD, sarcoidosis, etc).
* Presence of another chronic systemic inflammatory disease (rheumatoid arthritis or other connective-tissue disease, chronic infection such as osteomyelitis, inflammatory bowel disease, chronic active hepatitis, etc). Subjects with osteoarthritis, stable coronary artery disease, hypertension, or diabetes mellitus will not be excluded.
* Presence of malignant neoplasm within the last 3 years (with the exception of non-melanoma skin cancer).
* Clinically significant left or right ventricular dysfunction.
* Severe pulmonary hypertension (high blood pressure).
* Untreated obstructive sleep apnea:
* Subjects with a current diagnosis of sleep apnea not being treated with CPAP or BiPAP will be excluded.
* Subjects with a current diagnosis of sleep apnea being treated adequately (as determined by the investigators) will be included.
* Prader-Willi syndrome
* A known endocrinopathy causing obesity (e.g., Cushing's Syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-11; Primary Completion 2007-07 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Beuther, MD, Principal Investigator — National Jewish Medical and Research Center faculty
Locations (1):
- National Jewish Medical and Research Center, Denver, Colorado, United States